CLINICAL TRIAL: NCT03317379
Title: Evaluation of the Communities of Healing Mentorship/Support Group Program: Assessment of Preliminary Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Lisa Ranzenhofer, Assistant Professor of Clinical Psychology (in Psychiatry), New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7533
Record Dates: First submitted 2017-10-12; First posted 2017-10-23 (Actual); Results first posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Eating Disorder; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Intervention Model Description: Randomization occurs at the beginning of each individual's participation in the study. Participants are randomized to one condition and not re-randomized during any portion of the study
Masking Description: Since this is a behavioral intervention, participants, care providers, and investigators are aware of each patient's randomization. Outcomes are assessed electronically.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer mentorship (Experimental): Participants meet weekly with an adult peer mentor who has recovered from an eating disorder. The focus of meetings is on eating disorder symptoms and how to overcome them. The goal of this program is to reduce eating disorder symptoms directly by receiving support and guidance from someone who has been through it.
  Interventions: Behavioral: Peer mentorship; Behavioral: Recovery Record use with mentor
- Social support mentorship (Active Comparator): Participants meet weekly with an adult mentor who has not personally struggled with an eating disorder but who is dedicated to offering support. During weekly meetings, participants and mentors (and possibly 1-2 other mentees) engage in activities unrelated to the eating disorder. The goal of this program is to reduce eating disorder symptoms indirectly by exploring aspects of self outside the eating disorder.
  Interventions: Behavioral: Social support mentorship
- Wait list (No Intervention): Participants are on a wait list and then get matched with either type of mentor (of their choice) 6 months later

INTERVENTIONS:
Behavioral: Peer mentorship — Weekly meetings with a recovered peer mentor once per week. Dyads discuss eating disorder symptoms and how to overcome them.
  Arms: Peer mentorship
Behavioral: Social support mentorship — Weekly meetings with a social support mentor who has not personally struggled with an eating disorder, once per week. Dyads engage in activities unrelated to the eating disorder (e.g., a movie, a community event, volunteer work).
  Arms: Social support mentorship
Behavioral: Recovery Record use with mentor — Recovery Record is a smart phone or web-based application designed to provide recovery support to eating disorder patients. Includes a number of features aimed to promote recovery, such as a meal tracking, prompts for completing meals/snacks, tracking for additional symptoms such as stress and mood, motivational messages, information about coping strategies, and capacity to share logged data with clinicians and mentors.
  Arms: Peer mentorship

SUMMARY:
The goal of the study is to evaluate two 6-month adjunct interventions (peer mentorship and social support mentorship) for individuals with eating disorders. Individuals will be randomized to peer-mentorship, social support mentorship, or a wait-list and eating disorder symptoms will be evaluated at baseline and post-treatment.

DETAILED DESCRIPTION:
Eating disorders are serious mental illnesses associated with significant morbidity and high relapse rates. Patients are at especially high risk of relapse after leaving structured treatment (e.g., hospitalization). Adjunct interventions targeting patients' motivation and participation in treatment at these times may help patients recover from eating disorders. Project HEAL is a non-profit organization whose mission is to reduce suffering caused by eating disorders, and they have recently developed two adjunct, mentorship-based interventions for patients in recovery. In the peer mentorship condition, individuals meet weekly with a peer mentor who has previously recovered from an eating disorder in order to discuss symptoms and coping strategies. In the social support mentorship condition, individuals meet weekly with a social support mentor who has not personally struggled with an eating disorder in order to engage in activities unrelated to the eating disorder. The aim of the current study is to evaluate the feasibility and efficacy of this intervention. The design of the study is a three-arm randomized controlled trial comparing peer mentorship, social-support mentorship, and wait-list control conditions. Participants in the study will be randomized to one of the three conditions for six months. Wait-list participants will subsequently receive either type of mentorship. Participants will complete assessments of their eating disorder symptoms at baseline, monthly throughout the course of the study, and one year after beginning the study. Outcomes will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Current or past 6 months AN, BN, or BED
* Recent (within 6 months) discharge from structured treatment
* Involved in outpatient treatment at an appropriate level of care
* Medical stability
* Access to smart phone or computer to complete study assessments

Exclusion Criteria:

* Evidence of needing specialized treatment for another medical or mental health condition

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peer Mentorship | Social Support Mentorship | Wait List
Started | 20 | 18 | 22
Completed Intervention (Completed intervention defined as participated in intervention for at least 20 weeks (out of 6 months)) | 16 | 6 | 0
Completed (Completion defined as completion of at least one follow-up study interval) | 20 | 15 | 20
Not Completed | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer Mentorship | Social Support Mentorship | Wait List | Total
Number analyzed (Participants) | 20 | 18 | 22 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (7.6) | 31.0 (5.0) | 27.1 (7.5) | 28.5 (7.0)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Information about sex/gender for 1 participant in Social Support arm not reported due to privacy/confidentiality issue.
  Participants
    Female | 20 | 17 | 22 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 18 | 18 | 22 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 16 | 17 | 20 | 53
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index
Description: kg/m2
Time Frame: Baseline (month 0, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Population: Number of subjects with Anorexia Nervosa or Atypical Anorexia Nervosa (n =45). The number of participants with AN or Atypical AN is less than the total sample.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Peer Mentorship | Social Support Mentorship | Wait List
Number analyzed (Participants) | 15 | 14 | 16
kg/m2
  Baseline (month 0) | 21.9 (3.6) | 20.7 (2.7) | 21.5 (4.0)
  Month 1: number analyzed (Participants) | 12 | 9 | 14
  Month 1 | 21.9 (4.0) | 21.1 (2.8) | 21.5 (4.5)
  Month 2: number analyzed (Participants) | 12 | 6 | 7
  Month 2 | 22.6 (3.8) | 21.4 (3.3) | 21.6 (4.9)
  Month 3: number analyzed (Participants) | 10 | 6 | 5
  Month 3 | 21.6 (4.1) | 21.6 (4.1) | 21.7 (3.7)
  Month 4: number analyzed (Participants) | 8 | 5 | 8
  Month 4 | 21.3 (3.5) | 21.3 (3.5) | 24.4 (3.4)
  Month 5: number analyzed (Participants) | 10 | 3 | 8
  Month 5 | 21.8 (4.2) | 21.8 (4.2) | 23.5 (3.4)
  Month 6: number analyzed (Participants) | 8 | 8 | 7
  Month 6 | 22.8 (4.3) | 22.8 (4.3) | 23.4 (4.1)
Statistical Analysis 1: Comparison: Peer Mentorship vs Wait List; Test type: Superiority; p = .80, Mixed Models Analysis — .05 is the a priori threshold for statistical significance; estimate of fixed effects = 0.03, 95% CI 2-sided [-0.17 to 0.22], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Peer Mentorship vs Social Support Mentorship; Test type: Superiority; p = .32, Mixed Models Analysis — .05 is the a priori threshold for statistical significance; estimate of fixed effects = 0.10, 95% CI 2-sided [-0.10 to 0.30], Standard Error of Mean 0.1

2. Primary Outcome: Binge Days
Description: Units on a scale from 0 - 4 ( 0 = 0 days; 1 = A few (1-2) days; 2 = About half (3-4) days; 4 = Most (5-6) days; 4 = All (7) days Range was 0 - 4
Time Frame: Baseline through Week 28
Population: Number of participants with BN or BED
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Peer Mentorship | Social Support Mentorship | Wait List
Number analyzed (Participants) | 5 | 4 | 6
units on a scale
  Baseline | 1.0 (0.7) | 1 (2) | 1.3 (1.0)
  Week 1: number analyzed (Participants) | 3 | 3 | 3
  Week 1 | 0.67 (.58) | 1.33 (2.3) | 1.0 (1.0)
  Week 2: number analyzed (Participants) | 4 | 3 | 6
  Week 2 | 1.25 (0.5) | .33 (.57) | 1.3 (1.4)
  Week 3: number analyzed (Participants) | 3 | 4 | 6
  Week 3 | 0.67 (0.58) | 1 (2) | .7 (.5)
  Week 4: number analyzed (Participants) | 1 | 2 | 6
  Week 4 | 1 (0) | 0 (0) | .8 (.8)
  Week 5 Week 5: number analyzed (Participants) | 4 | 3 | 5
  Week 5 Week 5 | 1.5 (1.0) | 1.3 (2.3) | 1.2 (.8)
  Week 6: number analyzed (Participants) | 3 | 2 | 6
  Week 6 | .67 (.58) | 0.5 (0.7) | 1.5 (.8)
  Week 7: number analyzed (Participants) | 2 | 3 | 3
  Week 7 | 0 (0) | 1.0 (1.7) | .3 (.6)
  Week 8: number analyzed (Participants) | 4 | 3 | 6
  Week 8 | 0.25 (0.50) | 1.3 (1.5) | 1.1 (1.3)
  Week 9: number analyzed (Participants) | 1 | 1 | 5
  Week 9 | 1 (0) | 2 (0) | .6 (.5)
  Week 10: number analyzed (Participants) | 1 | 1 | 4
  Week 10 | 1 (0) | 1 (0) | 1.0 (1.4)
  Week 11: number analyzed (Participants) | 2 | 2 | 4
  Week 11 | 0 (0) | 1 (0) | .8 (1.0)
  Week 12: number analyzed (Participants) | 2 | 1 | 4
  Week 12 | 0.50 (0.71) | 0 (0) | 1.8 (1.0)
  Week 13: number analyzed (Participants) | 1 | 1 | 6
  Week 13 | 1 (0) | 1 (0) | .7 (.7)
  Week 14: number analyzed (Participants) | 1 | 1 | 2
  Week 14 | 1 (0) | 0 (0) | 1.0 (1.4)
  Week 15: number analyzed (Participants) | 2 | 1 | 6
  Week 15 | 0 (0) | 1 (0) | 1.0 (0.9)
  Week 16: number analyzed (Participants) | 5 | 1 | 6
  Week 16 | .43 (.79) | 2 (0) | 0.7 (0.8)
  Week 17: number analyzed (Participants) | 2 | 1 | 3
  Week 17 | .5 (.7) | 2 (0) | 1.0 (1.0)
  Week 18: number analyzed (Participants) | 1 | 1 | 6
  Week 18 | 1 (0) | 1 (0) | 1.4 (1.2)
  Week 19: number analyzed (Participants) | 1 | 1 | 4
  Week 19 | 0 (0) | 0 (0) | 1.0 (1.4)
  Week 20: number analyzed (Participants) | 1 | 1 | 5
  Week 20 | 1 (0) | 0 (0) | 1.2 (1.3)
  Week 21: number analyzed (Participants) | 2 | 1 | 6
  Week 21 | 1 (0) | 0 (0) | 1.3 (1.0)
  Week 22: number analyzed (Participants) | 1 | 1 | 6
  Week 22 | 1 (0) | 3 (0) | 0.9 (0.7)
  Week 23: number analyzed (Participants) | 1 | 1 | 4
  Week 23 | 0 (0) | 0 (0) | 1.8 (1.0)
  Week 24: number analyzed (Participants) | 1 | 0 | 6
  Week 24 | 1 (0) |  | 1.4 (1.4)
  Week 25: number analyzed (Participants) | 5 | 1 | 2
  Week 25 | 1 (0) | 3 (0) | 0 (0)
  Week 26: number analyzed (Participants) | 5 | 1 | 4
  Week 26 | .13 (.35) | 0 (0) | 1.3 (1.3)
Statistical Analysis 1: Comparison: Peer Mentorship vs Wait List; Test type: Superiority; p = 0.01, Mixed Models Analysis — .05 is the a priori threshold for statistical significance; estimate of fixed effects = .14, 95% CI 2-sided [0.03 to 0.24], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Peer Mentorship vs Social Support Mentorship; Test type: Superiority; p = 0.28, Mixed Models Analysis — .05 is the a priori threshold for statistical significance; estimate of fixed effects = 0.08, 95% CI 2-sided [-.07 to 0.23], Standard Error of Mean 0.07

3. Primary Outcome: Body Dissatisfaction Subscale of the Eating Disorder Symptom Inventory (EPSI)
Description: The Eating Pathology Symptoms Inventory (EPSI) is a self-report questionnaire that includes 8 subscales and we used the Body Dissatisfaction subscale. Each item is rated on a 5-point Likert-style scale (0 = Never; 4= Often) to describe how well each item describes the participant's experiences. Scores are derived by summing responses across the questions included in each subscale. The range for Body dissatisfaction is 0 - 28. Higher scores are reflective of greater eating pathology.
Time Frame: Baseline, Month 3, Month 6
Population: Not every person completed this measure at every time point.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Peer Mentorship | Social Support Mentorship | Wait List
Number analyzed (Participants) | 20 | 18 | 21
units on scale
  Baseline: number analyzed (Participants) | 20 | 13 | 21
  Baseline | 23.5 (4.3) | 19.9 (6.3) | 21.2 (8.0)
  Month 3: number analyzed (Participants) | 19 | 18 | 19
  Month 3 | 19.6 (6.9) | 19.4 (6.0) | 20.7 (6.1)
  Month 6: number analyzed (Participants) | 18 | 15 | 20
  Month 6 | 18.2 (7.5) | 21.2 (6.2) | 20.9 (6.5)
Statistical Analysis 1: Comparison: Peer Mentorship vs Wait List; Test type: Superiority; p = 0.03, Mixed Models Analysis — .05 is the a priori threshold for statistical significance; estimate of fixed effects = 0.61, 95% CI 2-sided [0.06 to 1.16], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Peer Mentorship vs Social Support Mentorship; Test type: Superiority; p = 0.02, Mixed Models Analysis; estimate of fixed effects = 0.68, 95% CI 2-sided [0.09 to 1.27], Standard Error of Mean 0.29

4. Primary Outcome: Cognitive Restraint Subscale of the Eating Disorder Symptom Inventory (EPSI)
Description: The Eating Pathology Symptoms Inventory (EPSI) is a self-report questionnaire that includes 8 subscales and we used the Cognitive Restraint subscale. Each item is rated on a 5-point Likert-style scale (0 = Never; 4= Often) to describe how well each item describes the participant's experiences. Scores are derived by summing responses across the questions included in each subscale. The range for Cognitive Restraint is 0 - 12. Higher scores are reflective of greater eating pathology.
Time Frame: Baseline, Month 3, Month 6
Population: Not every participant filled out this measure at every time point.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Peer Mentorship | Social Support Mentorship | Wait List
Number analyzed (Participants) | 20 | 18 | 21
units on scale
  Baseline | 7.1 (2.8) | 7.3 (3.0) | 7.1 (2.4)
  Month 3: number analyzed (Participants) | 19 | 13 | 19
  Month 3 | 6.2 (3.3) | 6.8 (3.0) | 7.3 (2.1)
  Month 6: number analyzed (Participants) | 18 | 15 | 20
  Month 6 | 5.6 (2.8) | 7.0 (2.7) | 7.4 (2.3)
Statistical Analysis 1: Comparison: Peer Mentorship vs Wait List; Test type: Superiority; p = 0.08, Mixed Models Analysis — .05 is the a priori threshold for statistical significance; estimate of fixed effects = 0.20, 95% CI 2-sided [-0.02 to 0.42], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Peer Mentorship vs Social Support Mentorship; Test type: Superiority; p = 0.12, Mixed Models Analysis — .05 is the a priori threshold for statistical significance; estimate of fixed effects = 0.18, 95% CI 2-sided [-0.04 to 0.41], Standard Error of Mean 0.12

5. Primary Outcome: Restricting Subscale of the Eating Disorder Symptom Inventory (EPSI)
Description: The Eating Pathology Symptoms Inventory (EPSI) is a self-report questionnaire that includes 8 subscales and we used the Restricting subscale. Each item is rated on a 5-point Likert-style scale (0 = Never; 4= Often) to describe how well each item describes the participant's experiences. Scores are derived by summing responses across the questions included in each subscale. The range for Restricting is 0 - 24. Higher scores are reflective of greater eating pathology.
Time Frame: Baseline, Month 3, Month 6
Population: Not every participant completed this measure at every timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peer Mentorship | Social Support Mentorship | Wait List
Number analyzed (Participants) | 20 | 18 | 21
units on a scale
  Baseline | 11.5 (7.2) | 10.8 (6.4) | 8.4 (4.6)
  Month 3: number analyzed (Participants) | 19 | 13 | 19
  Month 3 | 11.7 (6.6) | 10.6 (5.9) | 9.6 (4.9)
  Month 6: number analyzed (Participants) | 18 | 15 | 20
  Month 6 | 9.5 (6.1) | 10.2 (5.2) | 9.4 (4.9)
Statistical Analysis 1: Comparison: Peer Mentorship vs Wait List; Test type: Superiority; p = 0.18, Mixed Models Analysis — the a priori threshold for statistical significance was 0.05; estimate of fixed effects = .030, 95% CI 2-sided [-0.14 to 0.74], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Peer Mentorship vs Social Support Mentorship; Test type: Superiority; p = 0.50, Mixed Models Analysis — the a priori threshold for statistical significance was 0.05; estimate of fixed effects = 0.16, 95% CI 2-sided [-0.30 to 0.62], Standard Error of Mean 0.23

ADVERSE EVENTS:
Time Frame: Information about adverse events was collected throughout the 6-month randomized study period.
Description: Information about participants health status and health care utilization was collected as part of mid- and post-treatment outcome surveys. Additionally, participants could report an event to the study team or to their mentor, and these events were logged in the participants' chart and included in AE report.
Arm/Group | Peer Mentorship | Social Support Mentorship | Wait List
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/18 | 5/22
Other Adverse Events (participants affected / at risk) | 5/20 | 3/18 | 10/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Mentorship (N=20) | Social Support Mentorship (N=18) | Wait List (N=22)
Complication of spinal surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Pt had planned spinal surgery for which she was taken off blood thinner, and she then had a blood clot form in her leg, resulting in an inpatient hospitalization. She spent several days in the hospital and then recuperated at home.
Inpatient psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) — Two patients had psychiatric hospitalization for suicidal ideation
Medical hospitalization for medical instability due to anorexia nervosa (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) — Two patients were hospitalized for medical complications of anorexia nervosa and then treated for anorexia nervosa in an inpatient setting
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer Mentorship (N=20) | Social Support Mentorship (N=18) | Wait List (N=22)
Higher level of care for eating disorder (Psychiatric disorders) | 5 (5) | 3 (3) | 9 (11) — Higher level of care for eating disorder includes residential treatment, partial hospitalization/day program, or intensive outpatient treatment
Ankle injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Ankle injury of unknown type

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT03317379/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT03317379/SAP_001.pdf